CLINICAL TRIAL: NCT02460809
Title: Home-based tDCS and Hand Tracking Rehabilitation for Chronic Stroke
Brief Title: Home-based Non-invasive Brain Stimulation and Hand Tracking Rehabilitation for People With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Home tDCS
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- In-lab tDCS (Active Comparator): Three people with chronic stroke will participate in finger tracking training while receiving transcranial direct current stimulation (tDCS) in a controlled laboratory environment with an investigator.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- In-home tDCS (Experimental): Three people with chronic stroke will participate in finger tracking training while receiving transcranial direct current stimulation (tDCS) in their own home. Patients will be taught how to use a blue-tooth enabled telerehabilitation module that is being controlled by an investigator in the lab on the University campus. For safety, an investigator will be in the home with each patient during tDCS use and finger tracking training but will only be supervising procedures.
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation (tDCS) uses two surface electrodes placed on the scalp. These electrodes pass a low voltage current and modulate membrane potentials of underlying neurons.

SUMMARY:
This is a device feasibility study, which will assess telerehabilitation in people with chronic stroke using a combination of noninvasive brain stimulation and finger tracking training. Telerehabilitation allows patients to train in their own home which also allows for longer training periods than what is currently allowed clinically. Noninvasive transcranial direct current stimulation (tDCS) uses two surface electrodes connected to a small battery that will be attached to the head. This will be used to modulate neuronal excitability. With sensors attached to fingers and the wrist, the patient will move the joints to track a target displayed on a screen. The combined treatment will be applied in two experiments. The first will be on 3 patients coming to our lab and the second on 3 patients in their home, both under supervision. We will integrate the two components and test the resulting and novel treatment system for technical feasibility, which will set the stage for future efficacy studies under federal grant support. We hypothesize that the developed system will be safe and feasible.

DETAILED DESCRIPTION:
This study will assess the feasibility of a telerehabilitation protocol involving non-invasive brain stimulation. Therefore, the two arms of the study are 1) implementation of this protocol in a controlled laboratory setting and 2) implementation of this protocol in a patient's home, being set up by the patient but controlled remotely using a blue-tooth system by an investigator in a different location. The two arms of this study will occur successively with the first arm being completed with three patients followed by the second arm being completed with a second group of three patients.

ELIGIBILITY:
Inclusion Criteria:

* adult at least 18 years old
* stroke duration >6 months,
* Mini-Mental State Examination score 24 or higher
* presence of tactile sensation on the scalp
* at least 10 degrees of active finger or wrist motion in the stroke hand
* ability to walk 100 feet and transfer independently

Exclusion Criteria:

* seizure within past two years
* pregnancy
* metal inside the had (dental metal is permitted)
* implanted medical devices incompatible with tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Digit Span | First day of study and one day following the final treatment
  Short-term memory test using single numerical digits
Box and block | First day of study and one day following the final treatment
  Finger dexterity test using both paretic and nonparetic hands
Quantification of Compliance Questionnaire | First day of study and one day following the final treatment
User perception survey | First day of study and one day following the final treatment
  Survey

SECONDARY OUTCOMES:
Survey of symptoms questionnaire | Each day of study as well as one day following the final treatment

CONTACTS AND LOCATIONS:
Overall Officials: James Carey, PhD, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Van de Winckel A, Carey JR, Bisson TA, Hauschildt EC, Streib CD, Durfee WK. Home-based transcranial direct current stimulation plus tracking training therapy in people with stroke: an open-label feasibility study. J Neuroeng Rehabil. 2018 Sep 18;15(1):83. doi: 10.1186/s12984-018-0427-2. PMID 30227864